CLINICAL TRIAL: NCT06644365
Title: Examining the Effect of Acupressure Mat on Perceived Stress, Sleep Quality and Premenstrual Symptoms in Students Experiencing Premenstrual Syndrome: Randomized Controlled Study
Brief Title: Acupressure Mat on Perceived Stress, Sleep Quality and Premenstrual Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Sinem Ceylan, Asist. Prof., Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Premenstrual Symptoms; Effect of Acupressure Mat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Students will be given a placebo exercise on a flat yoga/exercise mat on the same days, in the same way and for the same duration as the intervention group.
  Interventions: Other: Basic mat
- intervention group (Experimental): They will be asked to lie on the acupressure mat for 15 minutes once a day, 3 days a week (Monday, Wednesday, Friday). A reminder message will be sent on the morning of the application so that participants do not forget and are motivated. After each application, participants will be asked to fill out the session monitoring chart.
  Interventions: Other: Acupresure mat

INTERVENTIONS:
Other: Acupresure mat — The Premenstrual Syndrome Scale will be applied and the scale results will be evaluated. Participants who score 132 and above on the scale will be considered to be experiencing PMS. The intervention will be made in the second phase of the study.This practice will continue for three menstrual cycles.
  Arms: intervention group
Other: Basic mat — The Premenstrual Syndrome Scale will be applied and the scale results will be evaluated. Participants who score 132 and above on the scale will be considered to be experiencing PMS. The intervention will be made in the second phase of the study.Participants in this group will also be sent a reminder message similar to the intervention group. This practice will continue for three menstrual cycles.
  Arms: control group

SUMMARY:
Purpose of the study: To examine the effect of acupressure mat on perceived stress, sleep quality and premenstrual symptoms in students with premenstrual syndrome.

Hypotheses of the study;

In the post-test and follow-up test between students who were applied acupressure mat and those who were applied plain mat;

H10: There is no difference in terms of severity of premenstrual symptoms.

H20: There is no difference in terms of perceived stress.

H30: There is no difference in terms of sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Using medication and/or non-medical methods to cope with PMS
* Having any gynecological disease (abnormal uterine bleeding, myoma, ovarian cyst, etc.)
* Using contraceptive medication.

Exclusion Criteria:

* Participants wanting to withdraw from the study at any stage of the study
* Participants not complying with the research plan
* Diagnosed with a psychiatric or gynecological disease during the study
* Participants starting to receive additional treatment for PMS during the study period

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Symptom Scale | just before the application starts (pre-test), 12 weeks after the application starts (after the application ends/post-test) and 16 weeks later (follow-up test).
  It was developed by Gençdoğan (2006) to measure the severity of premenstrual symptoms. The scale consists of 44 questions that measure the severity of premenstrual symptoms based on DSM-III and DSM-IV-R. It is a five-point Likert-type scale. In the scoring of the scale, the option "Never" is given 1 point, the option "Very little" is given 2 points, and the option "Sometimes" is given 3 points.
Perceived Stress Scale | just before the application starts (pre-test), 12 weeks after the application starts (after the application ends/post-test) and 16 weeks later (follow-up test).
  The scale was developed by Cohen et al. in 1983 to measure the stress a person perceives in a given situation and was adapted to Turkish by Eskin et al. (2013). The 5-point Likert-type scale (Never (0)-Very often (4)) contains a total of 14 items. 7 items with positive expressions are scored in reverse. The minimum score from 0 to a maximum of 56 points can be obtained from the scale. A high score indicates that the person is highly stressed.
Visual Analog Scale (VAS) Sleep Quality | just before the application starts (pre-test), 12 weeks after the application starts (after the application ends/post-test) and 16 weeks later (follow-up test).
  Students will be asked to evaluate their sleep quality with the Visual Analog Scale. VAS-sleep quality is a 10 cm long tool. "My sleep quality is very poor" is written on the left end of the scale and "My sleep quality is very good" is written on the right. A score of 10 from the scale indicates that sleep quality is high, while a score of 0 indicates that sleep quality is very poor.